CLINICAL TRIAL: NCT06373393
Title: SPIRIT: Study of the Patency of Spinal aRteries After the STABILISE Technique
Acronym: SPIRIT
Status: Enrolling by invitation | Type: Observational
Sponsor: Associacao para Investigacao e Desenvolvimento da Faculdade de Medicina - CETERA (Other)
Collaborators: Cardiovascular Center of the University of Lisbon (Unknown); Unidade Local de Saúde Santa Maria (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Aortic Dissection; Spinal Cord Ischemia
Keywords: aortic dissection; STABILISE; spinal cord ischemia; bare stent; stent-graft; endovascular repair
MeSH Terms: conditions — Aortic Dissection; Spinal Cord Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: STABILISE — STABILISE technique: "Stent assisted balloon induced intimal disruption and relamination in aortic dissection repair"

SUMMARY:
The aim of the study is to evaluate the impact of the stent-assisted balloon-induced intimal disruption and relamination in aortic dissection repair (STABILISE) technique in the patency of intercostal and lumbar arteries detectable on computed tomography angiography (CTA) in patients with type B aortic dissection and its correlation with the occurrence of spinal cord ischaemia (SCI).

Primary end-point: patency of the intercostal and lumbar arteries on follow-up CTA.

Secondary end-point: spinal cord ischaemia

DETAILED DESCRIPTION:
BACKGROUND AND STUDY INTRODUCTION

Endovascular treatment emerged over the last decade as the standard of care for complicated acute type B aortic dissection and the first step is usually the deployment of a thoracic endograft (TEVAR) aiming to cover the entry tear. TEVAR may be enough to fix malperfusion syndromes but is frequently associated with late aortic dilatation and unfavorable remodeling [1,2]. The failure of simple TEVAR to solve malperfusion syndromes led to the development of adjunctive techniques like direct stenting of the occluded arteries, fenestration of the lamella or the association of a self-expandable bare stent deployment across the visceral and renal arteries to increase the true lumen diameter and improve perfusion of those arteries.

The STABILISE technique to treat type B dissections is able to disrupt the lamella of the dissected aorta and consequently restore the uniluminal state of the aortic anatomy [3,4,5].

The dissection process is related to the detachment of the aortic side branch ostia (visceral, renal, iliacs, intercostals, lumbars) and therefore a potential status of malperfusion which is often related to severe clinical complications that should be properly managed. Additionally, when the lamella is brought back to the peripheral aortic wall, according to the STABILISE concept, the recovery of perfusion from the true lumen is unclear.

All these mechanisms, as well as the cover of the ostia of upper intercostal arteries by the stentgraft, may compromise the intercostal and lumbar arteries patency or the direct flow from the true lumen and therefore be related to the occurrence of spinal cord ischemia complications which prevalence was not yet determined [6-10].

FEASIBILITY AND PRELIMINARY DATA

Our research group carried out a pilot study, accepted for publication in the journal "Journal of Vascular Surgery Cases, Innovations and Techniques", on patency of intercostal arteries after treatment of type B aortic dissection with the STABILIZE technique. In this study, we observed a decrease in the permeability of the intercostal arteries in the area of the thoracic endoprosthesis, but we concluded that the permeability of the spinal arteries was not significantly affected by the coverage of the aorta with the uncovered stent nor by its aggressive ballooning to replace the intimal lamella. These findings constitute a step towards a better understanding of the safety of this technique.

STUDY DESIGN AND METHODS

This is a multi-center, non-randomized, retrospective observational analysis of patients treated with STABILISE technique for type B aortic dissection.

The following data will be collected:

* preoperative comorbidities.
* temporal phase of dissection (hyperacute, acute, subacute or chronic).
* procedural data (diameter and length of the stentgraft(s) and bare stent(s) and length of the covered aorta.
* occurrence of SCI at discharge and 30 days after procedure, according to the TARLOV scale.

Contrast-enhanced thoraco-abdominal CTA will be performed to patients pre-operatively and within 1 month, 6 months and yearly after the procedure.

Inclusion criteria

All patients with ≥ 18 years of age, with a type B dissection, treated according to the STABILISE technique

Exclusion criteria

- Aortic rupture.

CTA protocol Contrast-enhanced thoraco-abdominal CTA (with thin slices, preferably 1mm) will be performed to all patients pre-operatively and within 1 month, 6 months and then yearly after the procedure. Axial, coronal and column curvature based maximum intensity projections (MIP) with 10mm slice thickness will be performed and analyzed retrospectively.

After removing any patient's identification, the DICOM data will be sent, via WeTransfer, to the analysis center in Lisbon where the quantification and patency analysis will be performed.

Results evaluation The CTA images will be semi-quantitatively analyzed by two independent investigators and the number of visible intercostal and lumbar arteries in the stented aorta (stent-graft and dilated bare metal stent) will be evaluated.

The following parameters will be analyzed and reported in the attached sheet:

PRE-TREATMENT CTA

* Presence and patency of the intercostal and lumbar arteries specifying right and left sides.
* Origin of the intercostal and lumbar arteries - true lumen, false lumen (FL), both - specifying right and left sides

POST-TREATMENT CTA's

* Presence and patency of the intercostal and lumbar arteries (specifying right and left sides).
* Origin of the intercostal and lumbar arteries (TL, FL, both) in cases where the uniluminal state was not completely restored (specifying right and left sides).
* Patency of the distal portion of the intercostal and lumbar arteries when the ostium was covered by the stentgraft (specifying right and left sides).
* Patency of the intercostal and lumbar arteries in the area of the bare stent (specifying right and left sides).
* Patency of the intercostal and lumbar arteries in the area distal to the bare stent (specifying right and left sides).

All the assessed variables will be collected at the coordinating Center (Santa Maria Hospital), using the image data provided by the two participating centers.

ELIGIBILITY:
Inclusion Criteria:

* patients with type B dissection treated according to the STABILISE technique

Exclusion Criteria:

* Aortic rupture.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients with type B aortic dissection submitted to the STABILISE technique
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
number of patent intercostal and lumbar arteries | baseline (pre op) and 1, 6, 12 and 24 months after surgery
  number of patent intercostal and lumbar arteries after STABILISE

SECONDARY OUTCOMES:
number of patients with spinal cord ischemia | baseline (pre op) and 1month after surgery
  number of patients with spinal cord ischemia after STABILISE

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde Santa Maria, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No